CLINICAL TRIAL: NCT07073066
Title: Deep Cervical Lymphatic Venous Anastomosis in the Treatment of Alzheimer's Disease: A Multicenter, Prospective, Open-label, Blinded-Endpoint, Randomized Controlled Trial (CLEAN-AD)
Brief Title: Deep Cervical Lymphatic Venous Anastomosis in the Treatment of Alzheimer's Disease (CLEAN-AD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2025-089-02
Record Dates: First submitted 2025-05-11; First posted 2025-07-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Alzheimers Disease
Keywords: Alzheimers disease; Cervical Lymphatic Venous Anastomosis; Randomized Controlled Trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This multicenter, prospective, open-label, blinded-endpoint, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The intervention is performed by well-trained surgeons, and the endpoint assessment is evaluated blindly by well-trained neurologists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC-LVA treatment plus usual care (Experimental): The intervention requires to perform bilateral deep cervical lymphatic venous anastomosis (DC-LVA). The usual care includes patients who were not using or were currently using medications for improving cognitive function.
  Interventions: Procedure: DC-LVA treatment plus usual care
- Usual care (Active Comparator): The usual care group includes patients who were not using or were currently using medications for improving cognitive function.
  Interventions: Other: Usual care

INTERVENTIONS:
Procedure: DC-LVA treatment plus usual care — Through cervical incision, the deep cervical lymphatic tissue is anatomically dissected and anastomosed with the venous system of the neck. Under indocyanine green (ICG) navigation, the flow of lymphatic fluid into the vein could be observed via ICG tracing fluorescence after surgery.
  Other Names: LVA
  Arms: DC-LVA treatment plus usual care
Other: Usual care — The usual care group includes patients who were not using or were currently using medications for improving cognitive function.
  Arms: Usual care

SUMMARY:
This multicenter, prospective, open-label, blinded-endpoint, randomized controlled trial is to evaluate the efficacy and safety of deep cervical lymphatic venous anastomosis (DC-LVA) plus usual care versus usual care in reduing the score of clinical dementia rating-sum of boxes (CDR-SB) at 12 months in patients with moderate-to-severe Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a common neurodegenerative disorder affecting the elderly population. Global health data estimates that there are 50 million AD patients worldwide, and this number may triple to 150 million cases by 2050. Anti-amyloid β (Aβ) monoclonal antibodies have emerged as disease-modifying therapies for preclinical or mild AD, but the majority of candidate agents have failed to demonstrate clinical efficacy. For patients with moderate-to-severe AD, who comprise approximately 50% of the existing AD population, there are limitied treatment options in clinical practice. A series of case studies has suggested the efficacy of deep cervical lymphatic venous anastomosis (DC-LVA) in AD patients, however, there is currently no evidence from randomized controlled clinical trials.

The primary purpose of this study is to evaluate the efficacy and safety of deep cervical lymphatic venous anastomosis (DC-LVA) plus usual care versus usual care in reduing the score of clinical dementia rating-sum of boxes (CDR-SB) at 12 months in patients with moderate-to-severe Alzheimer's Disease (AD). This study also aims to assess the efficacy and safety of DC-LVA in reducing AD biomarker levels of brain Aβ PET imaging.

This trial is a multicenter, prospective, open-label, blinded-endpoint, randomized controlled trial. A total of 754 patients in 20 centers from China will be enrolled. Patients will be randomly assigned into DC-LVA plus usual care or usual care according to the ratio of 1:1. Face to face interviews will be made at baseline, 7 days (or hospital discharge), 3th months ± 7 days, 6th months ± 15 days, 9th months ± 15 days and 12th month ± 15 days after randomization. After 12 months, there will be 12 months open-label extension of follow-up, participants in the control group can choose to conduct DC-LVA. During the open-label extension phase, follow-up visits will be conducted every 3 months until 24th months after randomization.

Primary outcome is defined as the change of CDR-SB score at 12th months after randomization. The changes of CDR-SB score will be analyzed using a repeated measures mixed-effects model. Least squares means will be used to estimate the levels at each time point, and the mean difference with 95% confidence intervals will be calculated. Safety outcomes in the DC-LVA treatment group will be summarized using counts/percentages. Adverse events and serious adverse events will be summarized.

In exploratory outcome measures, the investigators will analyse the AD associated biomarkers in lymphatic tissue in the intervetnon group during the surgery, and analyse the change of fluid biomarkers ( AD associated biomarkers in peripheral blood, saliva, urine, and cerebrospinal fluid), the change of MRI brain volumes (total brain volume, hippocampal volume, lateral ventricle volume), the change of glymphatic function index(DTI-ALPS), the change of MRS metabolic markers (N-Acetylaspartate, Creatine, Choline, Lactate, Glutamate and Glutamine, myo-Inositol), and the change of artificial intelligence-assisted oculomotor/gait measurements during 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80 years, male or female.
2. Diagnosed with AD according to NIA-AA criteria.
3. Moderate-to-severe AD dementia, defined as Clinical Dementia Rating Scale Global Score (CDR-GS) ≥1.
4. Mini-Mental State Examination (MMSE) score 10-20.
5. The course of AD more than 6 months.
6. If receiving an approved AD treatment, must be on a stable drug dose for at least 3 months prior to Baseline. AD Treatment-naïve subjects can be entered into the study.
7. Have an identified caregiver (defined as a person able to support the subject for the duration of the study and who spends at least 8 hours per week with the subject). The caregiver must accompany with the participant at all study follow-up visits.
8. Signed informed consent (from the participant or their relative, and the caregiver).

Exclusion Criteria:

1. Any neurological condition other than AD that may affect cognitive function, including stroke, Parkinson's disease, epilepsy, intracranial tumors or space-occupying lesions, traumatic brain injury, intracranial infections, metabolic encephalopathy, etc.
2. Other causes of dementia, including vascular dementia, hereditary cerebral small vessel disease, vitamin deficiency, or any other etiology leading to dementia.
3. Previous evidence of severe stenosis (≥70%) in the middle cerebral artery and/or internal carotid artery.
4. Presence of primary psychiatric disorders (such as schizophrenia, schizoaffective disorder, major depressive disorder, or bipolar disorder) rather than psychiatric symptoms caused by AD.
5. Severe neurological deficits in limb movement, language, vision, hearing, or consciousness, or any condition that the investigator determines may prevent the completion of cognitive function assessments.
6. History of drug or alcohol abuse or dependence.
7. History of malignant tumors or prior radiotherapy or surgery involving the head and neck.
8. Major surgical procedures or severe head or body trauma within the past 30 days.
9. Presence of other life-threatening conditions with an expected survival time of less than 2 years.
10. Contraindications to head MRI (including cardiac pacemakers/defibrillators, ferromagnetic metal implants, etc.).
11. Severe diseases or functional impairment of the heart, lungs, liver, kidneys, or other solid organs, making the patient unable to tolerate anesthesia or DC-LVA.
12. Severe bleeding tendency (including but not limited to): platelet count <100×10⁹/L; heparin therapy within the last 48 hours with APTT ≥35 seconds; ongoing warfarin use with INR >1.7.
13. Requirement for long-term use of antithrombotic medications, with inability to discontinue them before surgery or potential risks associated with discontinuation.
14. Uncontrolled persistent hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure >95 mmHg).
15. Co-infection with HIV or Treponema pallidum, or any uncontrolled infectious disease.
16. Use of other investigational drugs or devices within 30 days prior to obtaining informed consent, or current participation in other interventional clinical studies.
17. Pregnancy, lactation, potential for pregnancy, or plans for pregnancy during the study period.
18. Immediate family members of the investigator (spouse, parents, children, or siblings), staff of the research institution or third-party organizations, or any other individuals with potential conflicts of interest related to the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
The change of Clinical Dementia Rating-Sum of Boxes score at 12th months after randomization | From baseline to 12th months after randomization
  The change of Clinical Dementia Rating-Sum of Boxes score (CDR-SB, 0-18 score, higher scores mean a worse outcome)

SECONDARY OUTCOMES:
The Change of Clinician's Interview-Based Impression of Change plus caregiver input score | From baseline to 12th months after randomization
  Clinician's Interview-Based Impression of Change plus caregiver input score (CIBIC-plus, 1-7 score, higher scores mean a worse outcome)
The Change of Neuropsychiatric Inventory Score | From baseline to 12th months after randomization
  Neuropsychiatric Inventory Score (NPI, 0-144 score, higher scores mean a worse outcome)
The Change of Aβ PET-CT Centiloid value | From baseline to 12th months after randomization
  The change of Aβ PET-CT Centiloid value at 12 months
The Change of Zarit Caregiver Interview of Alzheimer's Disease Score | From baseline to 12th months after randomization
  Zarit Caregiver Interview of Alzheimer's Disease Score (ZCI-AD, 0-88 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Assessment Scale-Activity of Daily Living score | From baseline to 12th months after randomization
  Alzheimer's Disease Assessment Scale-Activity of Daily Living score (ADCS-ADL, 0-78 score, higher scores mean a better outcome)
The Change of Mini-Mental State Examination Score | From baseline to 12th months after randomization
  Mini-Mental State Examination Score (MMSE, 0-30 score, higher scores mean a better outcome)
The Change of Clinical Dementia Rating-Sum of Boxes score | From baseline to 3th, 6th, 9th months after randomization
  Clinical Dementia Rating-Sum of Boxes score (CDR-SB, 0-18 score, higher scores mean a worse outcome
The Change of Clinician's Interview-Based Impression of Change plus caregiver input score | From baseline to 3th, 6th, 9th months after randomization
  Clinician's Interview-Based Impression of Change plus caregiver input score (CIBIC-plus, 1-7 score, higher scores mean a worse outcome)
The Change of Neuropsychiatric Inventory Score | From baseline to 3th, 6th, 9th months after randomization
  Neuropsychiatric Inventory Score (NPI, 0-144 score, higher scores mean a worse outcome)
The Change of Zarit Caregiver Interview of Alzheimer's Disease Score | From baseline to 3th, 6th, 9th months after randomization
  Zarit Caregiver Interview of Alzheimer's Disease Score (ZCI-AD, 0-88 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Assessment Scale-Activity of Daily Living score | From baseline to 3th, 6th, 9th months after randomization
  Alzheimer's Disease Assessment Scale-Activity of Daily Living score (ADCS-ADL, 0-78 score, higher scores mean a better outcome)
The Change of Mini-Mental State Examination Score | From baseline to 3th, 6th, 9th months after randomization
  Mini-Mental State Examination Score (MMSE, 0-30 score, higher scores mean a better outcome
The Change of Alzheimer's Disease Assessment Scale Cognitive Score | From baseline to 3th, 6th, 9th, 12th months after randomization
  Alzheimer's Disease Assessment Scale Cognitive score (ADCS-Cog-13, 0-85 score, higher scores mean a worse outcome)
The Change of Severe Impairment Batterty Score | From baseline to 3th, 6th, 9th, 12th months after randomization
  Severe Impairment Batterty Score (SIB, 0-100 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Composite Score | From baseline to 3th, 6th, 9th, 12th months after randomization
  Alzheimer's Disease Composite Score (ADCOMS, 0-1.97 score, higher scores mean a worse outcome) is calculated by a weighted items from three scales including ADCS-Cog, MMSE, and CDR-SB.

OTHER OUTCOMES:
The change of Clinical Dementia Rating-Sum of Boxes score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Clinical Dementia Rating-Sum of Boxes score (CDR-SB, 0-18 score, higher scores mean a worse outcome)
The Change of Clinician's Interview-Based Impression of Change plus caregiver input score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Clinician's Interview-Based Impression of Change plus caregiver input score (CIBIC-plus, 1-7 score, higher scores mean a worse outcome)
The Change of Neuropsychiatric Inventory Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Neuropsychiatric Inventory Score (NPI, 0-144 score, higher scores mean a worse outcome)
The Change of Zarit Caregiver Interview of Alzheimer's Disease Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Zarit Caregiver Interview of Alzheimer's Disease Score (ZCI-AD, 0-88 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Assessment Scale-Activity of Daily Living score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Alzheimer's Disease Assessment Scale-Activity of Daily Living score (ADCS-ADL, 0-78 score, higher scores mean a worse outcome)
The Change of Mini-Mental State Examination Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Mini-Mental State Examination Score (MMSE, 0-30 score, higher scores mean a better outcome)
The Change of Alzheimer's Disease Assessment Scale-Cognitive Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Alzheimer's Disease Assessment Scale-Cognitive Score (ADCS-Cog-13, 0-85 score, higher scores mean a worse outcome)
The Change of Severe Impairment Batterty Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Severe Impairment Batterty Score (SIB, 0-100 score, higher scores mean a worse outcome)
The Change of Alzheimer's Disease Composite Score during the open-label extension phase | From baseline to 15th, 18th, 21th, and 24th months after randomization
  Alzheimer's Disease Composite Score(ADCOMS, 0-1.97 score, higher scores mean a worse outcome) is calculated by a weighted items from three scales including ADCS-Cog, MMSE, and CDR-SB.
The incidence of perioperative complications in the intervention group within 7 days after randomization | From baseline to 7th days after randomization
  The incidence of perioperative complications in the intervention group

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hopital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No